CLINICAL TRIAL: NCT00299130
Title: A Randomized, Placebo Controlled, Double-blind, Parallel Group, International Study to Evaluate the Safety and Efficacy of Rituximab in Combination With Methotrexate, Compared to Methotrexate Monotherapy, in Patients With Active Rheumatoid Arthritis
Brief Title: A Study to Evaluate the Safety and Efficacy of Rituximab in Combination With Methotrexate Compared to Methotrexate Alone in Patients With Active Rheumatoid Arthritis
Acronym: SERENE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U2973g; WA17045 (Other: F. Hoffmann-La Roche)
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Results first posted 2013-06-28 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; Rituxan; SERENE
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Folic Acid; Methotrexate; Methylprednisolone; Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo + methotrexate (MTX) (Active Comparator): Participants received placebo intravenous infusion on Days 1 and 15. From Week 16 onwards, participants could switch to receive rituximab 0.5 g (on Days 1 and 15) every 24 weeks for up to 5 years if they were not in clinical remission and safety criteria were met. Placebo and rituximab infusions were preceded with 100 milligrams (mg) intravenous methylprednisolone. Participants also received a stable dose of 10-25 mg/week of MTX and ≥ 5 mg/week folic acid for the duration of their participation in the study.
  All participants entered a 48-week safety follow-up (SFU) period following the treatment period.
  Interventions: Drug: Folate; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Placebo; Drug: Rituximab
- Rituximab 2 x 0.5 g + MTX (Experimental): Participants received 0.5 g rituximab administered by intravenous infusion on Days 1 and 15. After Week 24, participants received further courses of rituximab every 24 weeks for up to 5 years if they were not in clinical remission and safety criteria were met. Rituximab infusions were preceded with 100 mg intravenous methylprednisolone.
  Participants also received a stable dose of 10-25 mg/week of methotrexate and ≥ 5 mg/week folic acid for the duration of their participation in the study.
  All participants entered a 48-week safety follow-up (SFU) period following the treatment period.
  Interventions: Drug: Folate; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Rituximab
- Rituximab 2 x 1.0 g + MTX (Experimental): Participants received 1.0 g rituximab administered by intravenous infusion on Days 1 and 15. After Week 24, participants received further courses of rituximab every 24 weeks for up to 5 years if they were not in clinical remission and safety criteria were met. Rituximab infusions were preceded with 100 mg intravenous methylprednisolone.
  Participants also received a stable dose of 10-25 mg/week of methotrexate and ≥ 5 mg/week folic acid for the duration of their participation in the study.
  All participants entered a 48-week safety follow-up (SFU) period following the treatment period.
  Interventions: Drug: Folate; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Rituximab

INTERVENTIONS:
Drug: Folate — A stable dose, ≥ 5 mg/week given as either a single dose or as a divided weekly dose, orally.
Drug: Methotrexate — A stable dose of between 10-25 mg/week, oral or parenteral, as prescribed by the treating physician.
Drug: Methylprednisolone — Intravenous infusion
Drug: Placebo — Placebo to rituximab intravenous infusion
  Arms: Placebo + methotrexate (MTX)
Drug: Rituximab — Intravenous infusion
  Other Names: MabThera®; Rituxan®

SUMMARY:
This study evaluated the efficacy and safety of rituximab in patients with active rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion criteria:

* Adult patients 18-80 years of age.
* Rheumatoid arthritis (RA) for ≥ 6 months, diagnosed according to the revised 1987 American College of Rheumatology (ACR) criteria for the classification of rheumatoid arthritis.
* Receiving outpatient treatment for RA.
* Swollen joint count (SJC) ≥ 8 (66 joint count), and tender joint count (TJC) ≥ 8 (68 joint count) at screening and baseline.
* At screening, either

  * C-reactive protein (CRP) ≥ 0.6 mg/dL (6 mg/L), or
  * Erythrocyte sedimentation rate (ESR) ≥ 28 mm/hour.
* Inadequate response to methotrexate, having received and tolerated at a dose of 10-25 mg/week it for ≥ 12 weeks.

Exclusion criteria:

* Rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA.
* Inflammatory joint disease other than RA, or other systemic autoimmune disorder.
* Diagnosis of juvenile rheumatoid arthritis, or RA before the age of 16.
* Surgery within 12 weeks of study or planned within 24 weeks of randomization.
* Previous treatment with any approved or investigational biological agent for RA, an anti-alpha4-integrin antibody or co-stimulation modulator, or cell-depleting therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.

REFERENCES:
- [Result] Emery P, Deodhar A, Rigby WF, Isaacs JD, Combe B, Racewicz AJ, Latinis K, Abud-Mendoza C, Szczepanski LJ, Roschmann RA, Chen A, Armstrong GK, Douglass W, Tyrrell H. Efficacy and safety of different doses and retreatment of rituximab: a randomised, placebo-controlled trial in patients who are biological naive with active rheumatoid arthritis and an inadequate response to methotrexate (Study Evaluating Rituximab's Efficacy in MTX iNadequate rEsponders (SERENE)). Ann Rheum Dis. 2010 Sep;69(9):1629-35. doi: 10.1136/ard.2009.119933. Epub 2010 May 20. PMID 20488885
- [Derived] Lal P, Su Z, Holweg CT, Silverman GJ, Schwartzman S, Kelman A, Read S, Spaniolo G, Monroe JG, Behrens TW, Townsend MJ. Inflammation and autoantibody markers identify rheumatoid arthritis patients with enhanced clinical benefit following rituximab treatment. Arthritis Rheum. 2011 Dec;63(12):3681-91. doi: 10.1002/art.30596. PMID 22127691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 511 participants were recruited and randomized between 27 Oct 2005 and 15 Nov 2006. Of these, 2 participants were randomized but received no infusions (one violated inclusion criteria and the other was randomized to rituximab 2 x 1.0 gram [g] + methotrexate [MTX] but failed to return). A total of 509 participants were treated.
Pre-assignment Details: Of the 509 participants, one participant was randomized first to rituximab 2 x 1.0 g + MTX and then to rituximab 2 x 0.5 g + MTX. No assessments were recorded or medication given after first randomization and all data used in analyses was following the second randomization; hence, participant is included only in rituximab 2 x 0.5 g + MTX arm.
Groups:
- Placebo + MTX: Participants received placebo intravenous infusion on Days 1 and 15. From Week 16 onwards, participants could switch to receive rituximab 0.5 g (on Days 1 and 15) every 24 weeks for up to 5 years if they were not in clinical remission and safety criteria were met. Placebo and rituximab infusions were preceded with 100 milligrams (mg) intravenous methylprednisolone. Participants also received a stable dose of 10-25 mg/week of MTX and ≥ 5 mg/week folic acid for the duration of their participation in the study.
  All participants entered a 48-week safety follow-up (SFU) period following the treatment period.
Period: Treatment Period (up to 5 Years)
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Started | 172 | 168 | 171
Treated | 172 (155 participants in placebo arm switched to active therapy (rituximab 2 x 0.5g) between Weeks 16-48.) | 167 | 170
Completed 24 Weeks | 159 | 162 | 166
Completed 48 Weeks | 155 | 157 | 158
Completed 144 Weeks | 133 | 138 | 132
Completed | 119 | 125 | 121
Not Completed | 53 | 43 | 50
Not completed — Adverse Event | 13 | 8 | 13
Not completed — Death | 1 | 3 | 1
Not completed — Insufficient Therapeutic Response | 19 | 6 | 6
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Refused Treatment | 12 | 12 | 19
Not completed — Failure to Return | 4 | 6 | 6
Not completed — Reason not Specified | 4 | 6 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 1
Period: Safety Follow-up (SFU) (48 Weeks)
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Started | 167 | 165 | 168
Completed | 122 | 120 | 123
Not Completed | 45 | 45 | 45
Not completed — Administrative/Other | 4 | 9 | 4
Not completed — Death | 4 | 5 | 3
Not completed — Did not Co-operate | 1 | 1 | 2
Not completed — Failure to Return | 14 | 7 | 15
Not completed — No SFU Week 48 Date Recorded | 0 | 1 | 0
Not completed — Withdrawal by Subject | 22 | 22 | 21
Period: Extended SFU (ESFU) (up to 5.1 Years)
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Started | 0 | 82 | 44
Completed | 0 | 74 | 38
Not Completed | 0 | 8 | 6
Not completed — Death | 0 | 3 | 0
Not completed — Failure to Return | 0 | 2 | 2
Not completed — Did not Cooperate/Withdrew Consent | 0 | 3 | 4

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received any part of an infusion.
Groups:
- Placebo + MTX: Participants received placebo intravenous infusion on Days 1 and 15. From Week 16 onwards, participants could switch to receive rituximab 0.5 g (on Days 1 and 15) every 24 weeks for up to 5 years if they were not in clinical remission and safety criteria were met. Placebo and rituximab infusions were preceded with 100 mg intravenous methylprednisolone. Participants also received a stable dose of 10-25 mg/week of MTX and ≥ 5 mg/week folic acid for the duration of their participation in the study.
  All participants entered a 48-week safety follow-up (SFU) period following the treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX | Total
Number analyzed (Participants) | 172 | 167 | 170 | 509
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.16 (12.39) | 51.91 (12.93) | 51.30 (12.64) | 51.80 (12.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 133 | 138 | 418
  Male | 25 | 34 | 32 | 91

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 20 Response at Week 24
Description: To achieve an ACR20 required at least a 20% improvement compared with Baseline in both tender joint counts (68 joints assessed for tenderness) and swollen joint counts (66 joints assessed for swelling), as well as a 20% improvement in three of the following five additional measurements:
  * Physician's global assessment of disease activity (assessed using a 100 mm Visual Analog Scale [VAS]);
  * Patient's global assessment of disease activity (assessed using a 100 mm VAS);
  * Patient's assessment of pain (assessed using a 100 mm VAS);
  * Health Assessment Questionnaire (HAQ; a patient completed questionnaire consisting of 20 questions, scored from 0-3);
  * Acute phase reactant: C-reactive protein (CRP) or, if CRP was missing, erythrocyte sedimentation rate (ESR).
  Participants who withdrew prematurely from the study prior to Week 24, who received rescue therapy or had insufficient data in order to calculate a clinical response were considered to be non-responders.
Time Frame: Baseline and Week 24
Population: Intent to treat population included all randomized participants who received at least 1 or part of an infusion. ACR was calculated using the last observation carried forward (LOCF) values for each component. Participants who withdrew prior to week 24, received rescue therapy or had insufficient data to calculate ACR were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percentage of participants | 23.3 | 54.5 | 50.6

2. Secondary Outcome: Percentage of Participants With an ACR50 Response at Week 24
Description: To achieve an ACR50 required at least a 50% improvement compared with Baseline in both tender joint counts (68 joints assessed for tenderness) and swollen joint counts (66 joints assessed for swelling), as well as a 50% improvement in three of the following five additional measurements:
  * Physician's global assessment of disease activity (assessed using a 100 mm Visual Analog Scale [VAS]);
  * Patient's global assessment of disease activity (assessed using a 100 mm VAS);
  * Patient's assessment of pain (assessed using a 100 mm VAS);
  * Health Assessment Questionnaire (HAQ; a patient completed questionnaire consisting of 20 questions, scored from 0-3);
  * Acute phase reactant: C-reactive protein (CRP) or, if CRP was missing, erythrocyte sedimentation rate (ESR).
  Participants who withdrew prematurely from the study prior to Week 24, who received rescue therapy or had insufficient data in order to calculate a clinical response were considered to be non-responders.
Time Frame: Baseline and Week 24
Population: Intent to treat population. ACR was calculated using LOCF values for each component. Participants who withdrew prior to Week 24, received rescue therapy or had insufficient data to calculate ACR were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percentage of participants | 9.3 | 26.3 | 25.9

3. Secondary Outcome: Percentage of Participants With an ACR70 Response at Week 24
Description: To achieve an ACR70 required at least a 70% improvement compared with Baseline in both tender joint counts (68 joints assessed for tenderness) and swollen joint counts (66 joints assessed for swelling), as well as a 70% improvement in three of the following five additional measurements:
  * Physician's global assessment of disease activity (assessed using a 100 mm Visual Analog Scale [VAS]);
  * Patient's global assessment of disease activity (assessed using a 100 mm VAS);
  * Patient's assessment of pain (assessed using a 100 mm VAS);
  * Health Assessment Questionnaire (HAQ; a patient completed questionnaire consisting of 20 questions, scored from 0-3);
  * Acute phase reactant: C-reactive protein (CRP) or, if CRP was missing, erythrocyte sedimentation rate (ESR).
  Participants who withdrew prematurely from the study prior to Week 24, who received rescue therapy or had insufficient data in order to calculate a clinical response were considered to be non-responders.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percentage of participants | 5.2 | 9.0 | 10.0

4. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS28-ESR) at Week 24
Description: The DAS28 is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables:
  * The number of swollen and tender joints assessed using the 28-joint count;
  * Erythrocyte sedimentation rate (ESR);
  * Patient's global assessment of disease activity measured on a 100 mm visual analog scale.
  The DAS28 score ranges from zero to ten. A DAS28 score above 5.1 means high disease activity whereas a DAS28 less than or equal to 3.2 indicates low disease activity. Remission is achieved by a DAS28 lower than 2.6.
Time Frame: Baseline and Week 24
Population: Intent to treat population with available data. DAS28 was calculated using last observation carried forward values for each of the component variables. If any of the components were missing then the DAS28 value will be missing.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 171 | 166 | 168
scores on a scale | -0.76 (1.304) | -1.71 (1.334) | -1.68 (1.342)

5. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response at Week 24
Description: A EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS28 score. The DAS28 score ranges from 0-10, with higher scores indicating more disease activity.
  A Good Response is defined as an improvement (decrease) in the DAS28 of more than 1.2 compared with Baseline and attainment of a DAS28 score of less than or equal to 3.2.
  A Moderate Response is defined as either:
  * an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 from Baseline and attainment of a DAS28 score of less than or equal to 5.1 or,
  * an improvement (decrease) in the DAS28 of more than 1.2 from Baseline and attainment of a DAS28 score of greater than 3.2.
  No Response is defined as either an improvement (decrease) in the DAS28 of less than or equal to 0.6, or an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 of more than 5.1.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population. LOCF was used for the individual components of the DAS-28. Non-responder imputation was used. Participants who withdrew prior to Week 24, who received rescue therapy or had insufficient data in order to calculate a EULAR response were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percentage of participants
  No Response | 66.3 | 33.5 | 37.1
  Moderate Response | 29.1 | 49.1 | 51.2
  Good Response | 4.7 | 17.4 | 11.8

6. Secondary Outcome: Percent Change From Baseline in Swollen Joint Count
Description: Sixty-six joints were assessed and classified as swollen/not swollen by pressure and joint manipulation on physical examination.
  The percentage change from baseline at each post-baseline visit was calculated as:
  [(post-baseline value minus baseline value) divided by Baseline value]*100.
  A negative percentage change from baseline score indicates an improvement.
Time Frame: Baseline, Week 24 and Week 48
Population: Intent-to-treat population, LOCF was used. "N" indicates the number of participants with non-missing data at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percent change
  Week 24 [N=172, 166, 170] | -21.6 (65.82) | -47.4 (43.49) | -49.1 (38.59)
  Week 48 [N=172, 166, 170] | -38.9 (66.83) | -54.0 (38.66) | -59.3 (37.04)

7. Secondary Outcome: Percent Change From Baseline in Tender Joint Count
Description: Sixty-eight joints were assessed and classified as tender/not tender by pressure and joint manipulation on physical examination.
  The percentage change from baseline at each post-baseline visit was calculated as:
  [(post-baseline value minus baseline value) divided by Baseline value]*100.
  A negative percentage change from baseline score indicates an improvement.
Time Frame: Baseline, Week 24 and Week 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percent change
  Week 24 [N=172, 166, 170] | -14.2 (69.20) | -42.5 (64.41) | -31.5 (66.52)
  Week 48 [N=172, 166, 170] | -37.1 (55.08) | -50.2 (62.74) | -45.1 (62.64)

8. Secondary Outcome: Percent Change From Baseline in Patient's Global Assessment of Disease Activity
Description: The participant's overall assessment of their current disease activity measured on a 100 mm horizontal visual analog scale (VAS). The left-hand extreme of the line (0 mm) was described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme (100 mm) as "maximum disease activity" (maximum arthritis disease activity).
  The percentage change from baseline at each post-baseline visit was calculated as:
  [(post-baseline value minus baseline value) divided by Baseline value]*100.
  A negative percentage change from baseline score indicates an improvement.
Time Frame: Baseline, Week 24 and Week 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percent change
  Week 24 [N=171, 166, 169] | -14.0 (48.94) | -31.5 (46.40) | -29.1 (54.43)
  Week 48 [N=171, 166, 169] | -28.0 (50.78) | -39.7 (40.53) | -36.6 (47.60)

9. Secondary Outcome: Percent Change From Baseline in Patient's Pain Assessment
Description: The participant's assessment of their current level of pain on a 100 mm horizontal visual analog scale (VAS), where the left-hand extreme of the line (0 mm) was described as "no pain" and the right-hand extreme (100 mm) as "unbearable pain".
  The percentage change from baseline at each post-baseline visit was calculated as:
  [(post-baseline value minus baseline value) divided by Baseline value]*100.
  A negative percentage change from baseline score indicates an improvement.
Time Frame: Baseline, Week 24 and Week 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percent change
  Week 24 [N=171, 166, 169] | -9.7 (52.58) | -25.7 (58.52) | -29.1 (53.11)
  Week 48 [N=171, 166, 169] | -24.4 (60.22) | -35.5 (50.45) | -36.3 (47.87)

10. Secondary Outcome: Percent Change From Baseline in Physician's Global Assessment of Disease Activity
Description: The physician's assessment of the participant's current disease activity on a 100 mm horizontal VAS, where the left-hand extreme of the line (0 mm) was described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme (100 mm) as "maximum disease activity".
  The percentage change from baseline at each post-baseline visit was calculated as:
  [(post-baseline value minus baseline value) divided by Baseline value]*100.
  A negative percentage change from baseline score indicates an improvement.
Time Frame: Baseline, Week 24 and Week 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percent change
  Week 24 [N=172, 166, 170] | -25.3 (38.52) | -36.9 (61.26) | -35.4 (46.99)
  Week 48 [N=172, 166, 170] | -39.4 (39.95) | -40.5 (74.54) | -49.0 (40.01)

11. Secondary Outcome: Percent Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score
Description: The Stanford Health Assessment Questionnaire disability index is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants choose from four response categories, ranging from 'without any difficulty' (Score=0) to 'unable to do' (Score=3). The overall score is the average of each of the 8 category scores and ranges from 0 to 3, where zero represents no disability and three very severe, high-dependency disability.
  The percentage change from baseline at each post-baseline visit was calculated as:
  [(post-baseline value minus baseline value) divided by Baseline value]*100.
  A negative percentage change from baseline score indicates an improvement.
Time Frame: Baseline, Week 24 and Week 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percent change
  Week 24 [N=172, 165, 170] | -14.7 (38.41) | -26.9 (40.89) | -23.4 (49.52)
  Week 48 [N=172, 165, 170] | -22.6 (39.63) | -30.2 (41.64) | -30.6 (39.95)

12. Secondary Outcome: Percent Change From Baseline in C-Reactive Protein
Description: C-Reactive Protein (CRP) was measured from blood samples by a central laboratory as a marker for inflammation.
  The percentage change from baseline at each post-baseline visit was calculated as:
  [(post-baseline value minus baseline value) divided by Baseline value]*100.
  A negative percentage change from baseline score indicates an improvement.
Time Frame: Baseline, Week 24 and Week 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percent change
  Week 24 [N=172, 166, 170] | 58.1 (385.23) | -27.5 (84.36) | -23.1 (119.75)
  Week 48 [N=172, 166, 170] | 40.1 (402.67) | -37.3 (94.65) | -34.9 (82.40)

13. Secondary Outcome: Percent Change From Baseline in Erythrocyte Sedimentation Rate
Description: Erythrocyte sedimentation rate (ESR) indirectly measures how much inflammation is in the body. A higher ESR is indicative of increased inflammation.
  The percentage change from baseline at each post-baseline visit was calculated as:
  [(post-baseline value minus baseline value) divided by Baseline value]*100.
  A negative percentage change from baseline score indicates an improvement.
Time Frame: Baseline, Week 24 and Week 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percent change
  Week 24 [N=172, 166, 169] | 8.0 (130.71) | -28.0 (42.20) | -29.2 (52.32)
  Week 48 [N=172, 166, 169] | -14.5 (68.55) | -31.3 (49.72) | -36.7 (51.49)

14. Secondary Outcome: Percent Change From Baseline in Short Form 36 Health Survey (SF-36) Summary Scores (Physical and Mental Components)
Description: The SF-36 measures the impact of disease on overall quality of life and consists of 36 questions split into two major components: physical health and mental health. Under physical health are the following four domains: physical health, bodily pain, physical functioning and physical role limitations. Under the mental health domain there are four domains; mental health, vitality, social functioning, and emotional role limitation. The individual domain scores are aggregated to derive a physical-component summary score and a mental-component summary score which range from 0 to 100, with higher scores indicating a better level of functioning.
  The percentage change from baseline at each post-baseline visit was calculated as:
  [(post-baseline value minus baseline value) divided by Baseline value]*100.
  A positive percentage change from baseline score indicates an improvement.
Time Frame: Baseline, Week 24 and Week 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percent change
  Physical Component: Week 24 [N=147, 152, 155] | 11.1 (27.63) | 23.7 (31.63) | 22.8 (33.09)
  Physical Component: Week 48 [N=154, 154, 162] | 21.3 (30.99) | 26.4 (35.81) | 27.4 (31.93)
  Mental Component: Week 24 [N=147, 152, 155] | 8.4 (29.43) | 12.6 (29.13) | 19.6 (56.64)
  Mental Component: Week 48 [N=154, 154, 162] | 12.7 (30.52) | 18.4 (38.87) | 18.7 (57.34)

15. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36) General Health Domain Score
Description: The SF-36 measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). The individual domain scores are calculated and transformed to range from 0 to 100, with higher scores indicating a better level of functioning.
  A positive change from baseline score indicates an improvement.
Time Frame: Baseline, Week 24 and Week 48
Population: Intent-to-treat population. "N" indicates the number of participants with non-missing data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
scores on a scale
  Week 24 [N=138, 154, 155] | 2.078 (7.3032) | 3.532 (8.2747) | 3.866 (9.2154)
  Week 48 [N=137, 148, 147] | 4.214 (8.2352) | 4.165 (9.5894) | 4.362 (8.1242)

16. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36) Bodily Pain Domain Score
Description: as for outcome 15
Time Frame: Baseline, Week 24 and Week 48
Population: Intent-to-treat population. "N" indicates the number of participants with non-missing data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
scores on a scale
  Week 24 [N=138, 152, 156] | 3.304 (8.5631) | 6.931 (8.2254) | 7.604 (8.5238)
  Week 48 [N=137, 147, 147] | 8.449 (9.3543) | 8.079 (9.5435) | 8.964 (8.9890)

17. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36) Physical Functioning Domain Score
Description: as for outcome 15
Time Frame: Baseline, Week 24 and Week 48
Population: Intent-to-treat population. "N" indicates the number of participants with non-missing data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
scores on a scale
  Week 24 [N=138, 154, 154] | 3.553 (8.4181) | 5.460 (8.3099) | 5.653 (9.6817)
  Week 48 [N=137, 148, 146] | 6.212 (9.6882) | 6.778 (8.7117) | 6.854 (9.3833)

18. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36) Physical Role Limitations Domain Score
Description: as for outcome 15
Time Frame: Baseline, Week 24 and Week 48
Population: Intent-to-treat population. "N" indicates the number of participants with non-missing data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
scores on a scale
  Week 24 [N=136, 153, 156] | 2.713 (8.7263) | 5.618 (9.0459) | 5.175 (8.8018)
  Week 48 [N=137, 148, 147] | 6.423 (9.6752) | 6.812 (9.8633) | 6.497 (8.4820)

19. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36) Mental Health Domain Score
Description: as for outcome 15
Time Frame: Baseline, Week 24 and Week 48
Population: Intent-to-treat population. "N" indicates the number of participants with non-missing data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
scores on a scale
  Week 24 [N=137, 153, 156] | 3.278 (8.6850) | 2.770 (9.9943) | 4.486 (9.4930)
  Week 48 [N=135, 147, 147] | 3.890 (8.7493) | 4.583 (10.5625) | 4.224 (9.9831)

20. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36) Vitality Domain Score
Description: as for outcome 15
Time Frame: Baseline, Week 24 and Week 48
Population: Intent-to-treat population. "N" indicates the number of participants with non-missing data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
scores on a scale
  Week 24 [N=137, 154, 156] | 3.631 (8.7662) | 4.230 (9.3631) | 5.910 (9.5802)
  Week 48 [N=135, 147, 147] | 6.853 (9.8221) | 5.925 (10.1495) | 5.869 (9.6168)

21. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36) Social Functioning Domain Score
Description: as for outcome 15
Time Frame: Baseline, Week 24 and Week 48
Population: Intent-to-treat population. "N" indicates the number of participants with non-missing data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
scores on a scale
  Week 24 [N=138, 154, 156] | 2.529 (9.6435) | 5.985 (10.2986) | 6.468 (10.8868)
  Week 48 [N=137, 148, 147] | 6.569 (10.6674) | 7.112 (11.5329) | 6.159 (11.0244)

22. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36) Emotional Role Limitations Domain Score
Description: as for outcome 15
Time Frame: Baseline, Week 24 and Week 48
Population: Intent-to-treat population. "N" indicates the number of participants with non-missing data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
scores on a scale
  Week 24 [N=136, 151, 155] | 1.829 (11.5405) | 4.634 (11.6419) | 4.464 (13.6883)
  Week 48 [N=137, 146, 146] | 4.724 (12.2649) | 6.257 (12.9640) | 4.446 (13.4036)

23. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Scores
Description: The FACIT-Fatigue questionnaire is a self-administered patient questionnaire that consists of 13 questions designed to measure the degree of fatigue experienced by participants in the previous 7 days. Participants respond to the questions using a value in the range of 0 (not at all) to 4 (very much). The scale score is computed by summing the item scores, after reversing those items that are worded in the negative direction. The FACIT-Fatigue subscale score ranges from 0 to 52, where higher scores represent less fatigue.
  A positive change from baseline score indicates an improvement.
Time Frame: Baseline, Week 24 and Week 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
scores on a scale
  Week 24 [N=170, 165, 168] | 2.661 (9.5093) | 5.564 (9.7438) | 6.398 (10.2143)
  Week 48 [N=170, 165, 169] | 5.506 (10.9651) | 6.269 (9.7495) | 6.203 (9.7833)

24. Secondary Outcome: Percentage of Participants With DAS28-ESR Low Disease Activity Score and Clinical Remission at Week 24
Description: The DAS28 is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables:
  * The number of swollen and tender joints assessed using the 28-joint count;
  * Erythrocyte sedimentation rate (ESR);
  * Patient's global assessment of disease activity measured on a 100 mm visual analog scale.
  The DAS28 score ranges from zero to ten. DAS28 above 5.1 indicates high disease activity.
  Low disease activity is defined by a DAS28 score less than or equal to 3.2. Remission is defined by a DAS28 score less than 2.6.
Time Frame: Week 24
Population: Intent to treat population with available data. DAS28 was calculated using last observation carried forward values for each of the component variables. If any of the components were missing then the DAS28 value will be missing. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 166 | 170
percentage of participants
  Low Disease Activity | 4.7 | 17.5 | 12.4
  Clinical Remission | 2.3 | 9.6 | 9.4

25. Secondary Outcome: Percentage of Participants With HAQ-DI Improved, Unchanged or Worsened at Week 24
Description: The Stanford Health Assessment Questionnaire disability index is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants choose from four response categories, ranging from 'without any difficulty' (Score=0) to 'unable to do' (Score=3). The overall score is the average of each of the 8 category scores and ranges from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. A negative change from baseline score indicates an improvement.
  Improved HAQ-DI is defined as a change from Baseline score less than or equal to -0.22.
  An Unchanged HAQ-DI is defined as a change from Baseline score greater than -0.22 and less than 0.22.
  A worsened HAQ-DI score is defined as a change from Baseline score of greater than or equal to 0.22.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population including participants with available data. LOCF was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 165 | 170
percentage of participants
  Improved | 47.7 | 66.1 | 58.2
  No change | 32.6 | 23.6 | 32.4
  Worsened | 19.8 | 10.3 | 9.4

26. Secondary Outcome: Percentage of Participants With HAQ-DI Improved, Unchanged or Worsened at Week 48
Description: as for outcome 25
Time Frame: Baseline and Week 48
Population: Intent-to-treat population including participants with available data. LOCF was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 165 | 170
percentage of participants
  Improved | 54.7 | 73.3 | 68.8
  No change | 29.1 | 17.0 | 25.3
  Worsened | 16.3 | 9.7 | 5.9

27. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response at Week 48
Description: A EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS-28 score.
  A Good Response is defined as an improvement (decrease) in the DAS28 of more than 1.2 compared with Baseline and attainment of a DAS28 score less than or equal to 3.2.
  A Moderate Response is defined as either:
  * an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 score of less than or equal to 5.1 or,
  * an improvement (decrease) in the DAS28 of more than 1.2 and attainment of a DAS28 score of greater than 3.2.
  No Response is defined as either an improvement (decrease) in the DAS28 of less than or equal to 0.6, or an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 score of 5.1 or higher.
Time Frame: Baseline and Week 48
Population: Intent-to-treat population. LOCF was used for the individual components of the DAS-28. Non-responder imputation was used. Patients who withdrew prior to week 48, who received rescue therapy or had insufficient data in order to calculate a EULAR response were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percentage of participants
  No Response | 41.3 | 26.9 | 31.8
  Moderate Response | 41.9 | 53.3 | 47.6
  Good Response | 16.9 | 19.8 | 20.6

28. Secondary Outcome: Percentage of Participants With DAS28-ESR Low Disease Activity Score and Clinical Remission at Week 48
Description: as for outcome 24
Time Frame: Week 48
Population: Intent to treat population including participants with available data. DAS28 was calculated using last observation carried forward values for each of the component variables. If any of the components were missing then the DAS28 value will be missing.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 171 | 165 | 169
percentage of participants
  Low Disease Activity | 18.1 | 20.0 | 24.3
  Clinical Remission | 7.0 | 9.1 | 11.2

29. Secondary Outcome: Percentage of Participants With an ACR50 Response at Week 48
Description: To achieve an ACR50 required at least a 50% improvement compared with Baseline in both tender joint counts (68 joints assessed for tenderness) and swollen joint counts (66 joints assessed for swelling), as well as a 50% improvement in three of the following five additional measurements:
  * Physician's global assessment of disease activity (assessed using a 100 mm Visual Analog Scale [VAS]);
  * Patient's global assessment of disease activity (assessed using a 100 mm VAS);
  * Patient's assessment of pain (assessed using a 100 mm VAS);
  * Health Assessment Questionnaire (HAQ; a patient completed questionnaire consisting of 20 questions, scored from 0-3);
  * Acute phase reactant: C-reactive protein (CRP) or, if CRP was missing, erythrocyte sedimentation rate (ESR).
  Participants who withdrew prematurely from the study prior to week 48, who received rescue therapy or had insufficient data in order to calculate a clinical response were considered to be non-responders.
Time Frame: Baseline and Week 48
Population: Intent to treat population. ACR was calculated using LOCF values for each component. Participants who withdrew prior to Week 48, received rescue therapy or had insufficient data to calculate ACR were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percentage of participants | 18.6 | 32.9 | 34.1

30. Secondary Outcome: Percentage of Participants With an ACR70 Response at Week 48
Description: To achieve an ACR70 required at least a 70% improvement compared with baseline in both tender joint counts (68 joints assessed for tenderness) and swollen joint counts (66 joints assessed for swelling), as well as a 70% improvement in three of the following five additional measurements:
  * Physician's global assessment of disease activity (assessed using a 100 mm Visual Analog Scale [VAS]);
  * Patient's global assessment of disease activity (assessed using a 100 mm VAS);
  * Patient's assessment of pain (assessed using a 100 mm VAS);
  * Health Assessment Questionnaire (HAQ; a patient completed questionnaire consisting of 20 questions, scored from 0-3);
  * Acute phase reactant: C-reactive protein (CRP) or, if CRP was missing, erythrocyte sedimentation rate (ESR).
  Participants who withdrew prematurely from the study prior to Week 48, who received rescue therapy or had insufficient data in order to calculate a clinical response were considered to be non-responders.
Time Frame: Baseline and Week 48
Population: as for outcome 29
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 172 | 167 | 170
percentage of participants | 9.3 | 12.6 | 13.5

31. Post Hoc Outcome: Time to Repletion of Peripheral CD19+ B-cells
Description: Peripheral CD19+ B-cell repletion was defined as a CD19+ B-cell count that returned to the Baseline value or returned to ≥ the lower limit of normal, whichever was lower.
Time Frame: Beginning of the first infusion (Day 1) in the last treatment cycle until repletion or the end of the study (approximately 6.5 years)
Population: Extended safety follow-up population: All participants who were randomized, received any part of a rituximab infusion, and entered the extended safety follow-up period.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Rituximab 2 x 0.5 g + MTX | Rituximab 2 x 1.0 g + MTX
Number analyzed (Participants) | 80 | 43
Weeks | 110.3 [89.6 to 148.3] | 109.6 [94.1 to 134.9]

32. Post Hoc Outcome: Percentage of Participants With Low Immunoglobulin Concentrations Pre- and Post-Rituximab Treatment
Description: A low immunoglobulin concentration was defined as a concentration below the lower level of normal.
Time Frame: Baseline (pre-rituximab), Beginning of the safety follow-up period to the end of the study (approximately 6 years) (post-rituximab)
Population: Safety follow-up population: All participants who were randomized and received any part of a rituximab infusion. Number of participants analyzed = participants with available data. "N" indicates the number of participants with non-missing data at each time point.
Measure: Number; unit: Percentage of participants
Groups:
- Rituximab + MTX: Participants received 0.5 g or 1.0 g rituximab administered by intravenous infusion on Days 1 and 15. After Week 24, participants received further courses of rituximab every 24 weeks for up to 5 years if they were not in clinical remission and safety criteria were met. Rituximab infusions were preceded with 100 mg intravenous methylprednisolone.
  Participants also received a stable dose of 10-25 mg/week of methotrexate and ≥ 5 mg/week folic acid for the duration of their participation in the study.
  All participants entered a 48-week safety follow-up (SFU) period following the treatment period.
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 491
Percentage of participants
  Pre-Rituximab (N=490) | 0.2
  Post-Rituximab (N=491) | 5.1

ADVERSE EVENTS:
Time Frame: Up to 5.1 years after last dose in treatment period (treatment period = up to 5 years)
Description: During the 5-year treatment period, all adverse events (AEs) regardless of seriousness were reported. During the standard 48-week safety follow-up (SFU) and extended safety follow-up (ESFU), all serious adverse events (SAEs) and all non-serious infections were reported.
Groups:
- Placebo + MTX: Includes all data for participants who remained on placebo, and data up to the point of switch if the participant switched to treatment with rituximab.
  Participants received placebo intravenous infusion on Days 1 and 15. From Week 16 onwards, participants could switch to receive rituximab 0.5 g (on Days 1 and 15) every 24 weeks for up to 5 years if they were not in clinical remission and safety criteria were met. Placebo and rituximab infusions were preceded with 100 mg intravenous methylprednisolone. Participants also received a stable dose of 10-25 mg/week of MTX and ≥ 5 mg/week folic acid for the duration of their participation in the study.
  All participants entered a 48-week safety follow-up (SFU) period following the treatment period.
- Rituximab 1.0 g + MTX: Participants received 1.0 g rituximab administered by intravenous infusion on Days 1 and 15. After Week 24, participants received further courses of rituximab every 24 weeks for up to 5 years if they were not in clinical remission and safety criteria were met. Rituximab infusions were preceded with 100 mg intravenous methylprednisolone. Participants also received a stable dose of 10-25 mg/week of methotrexate and ≥ 5 mg/week folic acid for the duration of their participation in the study.
  All participants entered a 48-week safety follow-up (SFU) period following the treatment period.
- Switch Population: Placebo + MTX: Includes all data up to the point of switch for participants in the Placebo + Methotrexate treatment group who switched to treatment with rituximab after Week 24.
- Switch Population: Rituximab: Includes all data from the point of switch for participants who switched from Placebo + Methotrexate to treatment with rituximab.
- Rituximab 2 x 0.5 g + MTX - Extended Safety Follow-up Period; Rituximab 2 x 1.0 g + MTX - Extended Safety Follow-up Period: Participants received no treatment during the extended safety follow-up period.
Arm/Group | Placebo + MTX | Rituximab 2 x 0.5 g + MTX | Rituximab 1.0 g + MTX | Switch Population: Placebo + MTX | Switch Population: Rituximab | Rituximab 2 x 0.5 g + MTX - Extended Safety Follow-up Period | Rituximab 2 x 1.0 g + MTX - Extended Safety Follow-up Period
Serious Adverse Events (participants affected / at risk) | 16/172 | 52/167 | 46/170 | 12/155 | 45/155 | 8/82 | 2/44
Other Adverse Events (participants affected / at risk) | 112/172 | 149/167 | 151/170 | 99/155 | 131/155 | 5/82 | 2/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + MTX (N=172) | Rituximab 2 x 0.5 g + MTX (N=167) | Rituximab 1.0 g + MTX (N=170) | Switch Population: Placebo + MTX (N=155) | Switch Population: Rituximab (N=155) | Rituximab 2 x 0.5 g + MTX - Extended Safety Follow-up Period (N=82) | Rituximab 2 x 1.0 g + MTX - Extended Safety Follow-up Period (N=44)
Pneumonia (Infections and infestations) | 1 | 3 | 4 | 1 | 3 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 1 | 2 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 1 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abscess soft tissue (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tubo-ovarian abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 4 | 3 | 0 | 3 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Traumatic coma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 5 | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weaknes (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Femoral hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ileal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 3 | 1 | 2 | 3 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pleuropericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
T-cell prolymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 1 | 3 | 1 | 0
Demyelination (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Benign intracranial hypertension (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 2 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Testicular necrosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device failure (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fibrosis (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hernia obstructive (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intra-abdominal haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis B DNA increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo + MTX (N=172) | Rituximab 2 x 0.5 g + MTX (N=167) | Rituximab 1.0 g + MTX (N=170) | Switch Population: Placebo + MTX (N=155) | Switch Population: Rituximab (N=155) | Rituximab 2 x 0.5 g + MTX - Extended Safety Follow-up Period (N=82) | Rituximab 2 x 1.0 g + MTX - Extended Safety Follow-up Period (N=44)
Upper respiratory tract infection (Infections and infestations) | 13 | 59 | 50 | 13 | 39 | 0 | 0
Nasopharyngitis (Infections and infestations) | 17 | 43 | 42 | 16 | 34 | 0 | 0
Urinary tract infection (Infections and infestations) | 12 | 41 | 25 | 9 | 34 | 5 | 2
Bronchitis (Infections and infestations) | 3 | 27 | 25 | 2 | 24 | 0 | 0
Sinusitis (Infections and infestations) | 6 | 24 | 21 | 6 | 29 | 0 | 0
Gastroenteritis (Infections and infestations) | 8 | 15 | 14 | 7 | 17 | 0 | 0
Influenza (Infections and infestations) | 1 | 17 | 20 | 1 | 13 | 0 | 0
Pharyngitis (Infections and infestations) | 10 | 15 | 11 | 10 | 9 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 9 | 8 | 0 | 7 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 10 | 4 | 2 | 5 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 2 | 8 | 1 | 9 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 30 | 49 | 36 | 26 | 31 | 0/0 | 0/0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 22 | 14 | 3 | 10 | 0/0 | 0/0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 9 | 15 | 2 | 7 | 0/0 | 0/0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 8 | 10 | 1 | 8 | 0/0 | 0/0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 7 | 7 | 4 | 10 | 0/0 | 0/0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 9 | 9 | 1 | 7 | 0/0 | 0/0
Infusion related reaction (Injury, poisoning and procedural complications) | 33 | 59 | 59 | 28 | 39 | 0/0 | 0/0
Fall (Injury, poisoning and procedural complications) | 5 | 14 | 5 | 4 | 18 | 0/0 | 0/0
Laceration (Injury, poisoning and procedural complications) | 1 | 2 | 10 | 1 | 6 | 0/0 | 0/0
Diarrhoea (Gastrointestinal disorders) | 7 | 27 | 20 | 7 | 20 | 0/0 | 0/0
Nausea (Gastrointestinal disorders) | 4 | 21 | 17 | 4 | 12 | 0/0 | 0/0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 7 | 10 | 2 | 4 | 0/0 | 0/0
Dyspepsia (Gastrointestinal disorders) | 3 | 4 | 4 | 3 | 11 | 0/0 | 0/0
Headache (Nervous system disorders) | 6 | 18 | 15 | 5 | 16 | 0/0 | 0/0
Dizziness (Nervous system disorders) | 4 | 11 | 10 | 3 | 0 | 0/0 | 0/0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 13 | 22 | 7 | 11 | 0/0 | 0/0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 10 | 0 | 6 | 0/0 | 0/0
Hypertension (Vascular disorders) | 3 | 28 | 18 | 2 | 15 | 0/0 | 0/0
Fatigue (General disorders) | 1 | 13 | 11 | 0 | 8 | 0/0 | 0/0
Oedema peripheral (General disorders) | 2 | 9 | 12 | 2 | 5 | 0/0 | 0/0
Depression (Psychiatric disorders) | 0 | 15 | 7 | 0 | 7 | 0/0 | 0/0
Insomnia (Psychiatric disorders) | 7 | 9 | 8 | 6 | 5 | 0/0 | 0/0
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 13 | 6 | 3 | 7 | 0/0 | 0/0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 7 | 9 | 1 | 5 | 0/0 | 0/0
Rash (Skin and subcutaneous tissue disorders) | 1 | 9 | 7 | 1 | 6 | 0/0 | 0/0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 9 | 6 | 0 | 3 | 0/0 | 0/0
Anaemia (Blood and lymphatic system disorders) | 5 | 9 | 12 | 4 | 7 | 0/0 | 0/0
Hepatotoxicity (Hepatobiliary disorders) | 2 | 8 | 7 | 2 | 8 | 0/0 | 0/0
Vertigo (Ear and labyrinth disorders) | 2 | 8 | 6 | 2 | 9 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.